CLINICAL TRIAL: NCT05540483
Title: Disitamab Vedotin（RC-48 ）Combined With Zimberelizumab（GLS-010） in HER2-overexpressed Patients With Previously Treated Unresectable Biliary Tract Cancer，A Single-arm, Open-label, Phase II Clinical Trail（RIGHT Study）
Brief Title: RC-48 Combined With GLS-010 in HER2-overexpressed Patients With Previously Treated Unresectable Biliary Tract Cancer
Acronym: RIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Xiaofeng Chen, Associate chief physician, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Xiaofeng Chen
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Biliary Carcinoma
MeSH Terms: interventions — zimberelimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Disitamab Vedotin combined with Zimberelizumab
  Interventions: Drug: Disitamab Vedotin combined with Zimberelizumab

INTERVENTIONS:
Drug: Disitamab Vedotin combined with Zimberelizumab — Treatment regimen: Disitamab Vedotin , 2.5mg/kg, intravenously D1, once every 14 days (Q2W), combined with Zimberelizumab, 240mg, intravenously D1, once every 14 days (Q2W).
  Other Names: RC-48 combined with GLS-010

SUMMARY:
This is a multicenter, single-arm, open-labal, phase II clinical study with a planned enrollment of 31 patients with HER2-overexpressing unresectable locally advanced or metastatic biliary carcinoma who had failed previous treatment. The efficacy and safety of the study were evaluated according to RECIST V1.1.

DETAILED DESCRIPTION:
The study included a screening period, a treatment period, and a follow-up period.

Screening period: Subjects who are fully aware of the study and have signed an informed consent form should complete all screening procedures within 28 days before the first dose. Only eligible subjects can be enrolled in the study. Prior to enrollment, subjects should provide a test report confirming HER2 overexpression, defined in this study as IHC 2+ or 3+. Official reports from local hospitals or genetic testing companies are acceptable. All subjects provided adequate tumor tissue samples (archived or fresh biopsy samples) for evaluation and confirmation of HER2 expression and genetic testing (15 paraffin sections, 5-10um thick) before study administration. Considering the accessibility of clinical specimens, specimens are not mandatory.

Treatment period: Each treatment period was 14 days. Treatment regimen: Disitamab Vedotin, 2.5mg/kg, intravenously D1, once every 14 days (Q2W), combined with Zimberelizumab, 240mg, intravenously D1, once every 14 days (Q2W). Study treatment will be continued until the subject has an intolerable toxic effect, withdrawal of informed consent, and disease progression as confirmed by RECIST V1.1 (when the subject has disease progression as assessed by the investigator according to RECIST V1.1, the investigator will then assess whether the subject still has clinical benefit. If the subject is considered to have continued clinical benefit and meets the criteria for continuing treatment after disease progression, the subject may continue to receive the study drug; Treatment may be discontinued if the subject is no longer considered to have clinical benefit), or any other termination criteria specified in the protocol, whichever comes first. Within the time window specified in each cycle, the subject will complete a physical examination, laboratory tests, and other tests to assess the subject's safety. Imaging evaluations of tumors were performed every 6 weeks (42±3 days) during study treatment. Tumor evaluation must include all known lesions in the abdomen, pelvis, and other sites. Scans of suspected lesions and bone may be performed at the investigator's discretion. The assessment methods used throughout the study should be as similar as possible. The preferred method is enhanced computed tomography (CT) or magnetic resonance imaging (MRI).

Follow-up period: including safety follow-up and survival follow-up. At the end of treatment, all subjects will be followed up for safety until 28 days after the last dose. Subjects who discontinue treatment for reasons other than PD will be followed up at the planned frequency until PD occurs, consent is withdrawn, or follow-up is lost, whichever occurs first. After completion of treatment and safety follow-up, all subjects were followed for survival (OS data were collected every 3 months ±14 days) until death, withdrawal of informed consent, loss to follow-up, or termination of the study, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study and signed informed consent;
2. Age 18-75, regardless of gender;
3. Unresectable local advanced or metastatic biliary malignancies confirmed by histopathology or cytology, including intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma and gallbladder carcinoma, excluding ampullary carcinoma;
4. Prior to enrollment, provide test reports confirming HER2 overexpression (defined as an immunohistochemical IHC score of 2+ or 3+), and provide sufficient sections of tumor tissue samples (archived or fresh biopsy samples) to evaluate and confirm HER2 expression, as well as other biomarker tests; Considering the availability of clinical specimens, specimens are not mandatory;
5. Subjects who progressed after prior first-line or above systemic therapy, or who progressed during or within 6 months after completion of adjuvant therapy, may be selected;
6. AE of previous medication/medical intervention is required to have been restored to baseline or ≤ grade 1 (NCI-CTCAE V5.0), except for AE such as hair loss or fatigue that does not affect subsequent treatment;
7. Subject will have at least one measurable lesion as per RECIST V1.1. The measurable target lesions in CT or MRI were defined as: according to RECIST V1.1 standard, the measurable length diameter of lesions ≥10 mm or the short diameter of enlarged lymph nodes ≥15 mm; The lesions that have previously received local treatment can be used as targets if their progression is confirmed according to RECIST V1.1 criteria;
8. ECOG Score: 0-2;
9. Estimated survival ≥12 weeks;
10. The function of the main organs is good, that is, the relevant examination indexes within 7 days before study administration meet the following requirements:

    A) Routine blood test:

    i. Hemoglobin ≥90 g/L (no blood transfusion within 14 days); ii. Neutrophil count > 1.5×109/L; iii. Platelet count ≥80×109/L;

    B) Biochemical examination:

    i. Total bilirubin ≤2.5×ULN (upper limit of normal value); ii. Serum alanine aminotransferase (ALT) or AST ≤2.5×ULN; ALT or AST if intrahepatic invasion is present (such as iCCA or liver metastasis)5 x ULN or less; iii. Endogenous creatinine clearance ≥60 mL /min (Cockcroft-Gault formula); C) Cardiac Doppler ultrasound assessment: left ventricular ejection fraction (LVEF)≥50%; D) No obvious abnormality of myocardial enzyme profile;
11. If subject has active hepatitis B virus (HBV) infection: HBV-DEoxyribonucleic acid (DNA) must be < 1000 IU/ mL and willing to receive antiviral therapy throughout the study period;
12. For female subjects: surgically sterilized, postmenopausal, or have consented to use a medically approved contraceptive during study treatment and for 6 months after the study treatment period; Serum or urine pregnancy tests must be negative during the 7 days prior to study enrollment and must be non-lactation. Male subjects: patients who agreed to use a medically approved contraceptive during study treatment and for 6 months after the end of study treatment; For specific contraceptive measures and definitions of women of childbearing age, see Appendix 1 contraceptive Measures, definitions of women of childbearing age and contraceptive requirements.

Exclusion Criteria:

1. Participated in clinical trials of other drugs within 4 weeks prior to the start of study administration;
2. Prior treatment with antibody-conjugated drugs targeting HER2; Patients who had previously received trastuzumab, pertuzumab, pyrrolitinib and other anti-HER2 therapy were eligible; Patients who had previously received PD-1 mab could be included; Patients who have previously been treated with taxoid-based drugs need to be eluted for more than 2 weeks.
3. Known prior allergy to monoclonal antibodies or to any of the test drug components;
4. Past history of other active malignancies within the past 5 years. Complete remission of basal cell carcinoma of the skin, superficial bladder, squamous cell carcinoma of the skin, carcinoma of the prostate in situ, or carcinoma of the cervix in situ for at least 2 years as of the date of first administration of the study drug and no additional treatment is required or expected during the study period;
5. Subjects with active central nervous system (CNS) metastases. Subjects with a current history or evidence of meningeal metastasis. Subjects are eligible to participate if CNS metastases are adequately treated (surgery or radiation) and their neurological function returns to baseline (other than residual signs or symptoms associated with CNS treatment) for at least 2 weeks prior to enrollment;
6. Clinically significant or poorly controlled heart disease, such as a history of unstable angina; Patients who were newly diagnosed with angina pectoris within 3 months before screening or had myocardial infarction within 6 months before screening; Arrhythmias (including QTcF: ≥450 ms for men and ≥470 ms for women) requiring long-term use of antiarrhythmic drugs and New York Heart Association classification ≥II cardiac insufficiency;
7. Patients with severe exudation accompanied by clinical symptoms (such as massive pleural effusion, ascites or pericardial effusion) and requiring repeated therapeutic puncture and drainage (allowing the use of catheters) before the first drug administration in the study;
8. A history of human immunodeficiency virus infection or other acquired or congenital immunodeficiency disease, or a history of organ transplantation;
9. Severe infection, including but not limited to hospitalization for infection, bacteremia, or severe pneumonia complications, within 2 weeks prior to the start of study treatment; Oral or intravenous administration of therapeutic antibiotics within 1 week prior to initiation of study treatment (allowing prophylactic antibiotics, such as those to prevent urinary tract infections or exacerbations of chronic obstructive pulmonary disease, to qualify for study);
10. There is active autoimmune disease or a history of autoimmune disease and may recur (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, the pituitary gland inflammation, vasculitis, nephritis, thyroid function, thyroid function decrease [just by hormone replacement therapy can control subjects can be incorporated into]); Subjects with skin diseases that do not require systematic treatment, such as vitiligo and psoriasis, controlled type I diabetes treated with insulin, or asthma that has been completely resolved in childhood and does not require any intervention as adults may be included; Asthma patients requiring medical intervention with bronchodilators were excluded;
11. Subjects requiring systematic treatment with corticosteroids (>10 mg/ day equivalent of prednisone) or other immunosuppressants within 14 days prior to initial use of the study drug;
12. Live vaccines (e.g. influenza virus vaccine, human papillomavirus vaccine) should be administered within 4 weeks prior to treatment with the study drug, and all vaccines except inactive vaccines should not be used during treatment;
13. Pregnant or lactating women;
14. Exclude, in the investigator's judgment, other disease or laboratory evidence that may pose a serious threat to patient safety or is not in the best interest of patient participation (including but not limited to: Superior vena cava syndrome, severe lung disease [untreated TB, untreated or within 3 months before delivery for the first time in research and treatment of pulmonary embolism, active pneumonia] except obstructive pneumonia, poor control of epilepsy, mental illness or in the near future plans for organ transplant, has inherited or acquired bleeding tendency);
15. Exclude, at the investigator's discretion, other conditions that might confuse the study results or affect the subjects' ability to follow the study procedures, such as alcoholism, drug abuse, mental disorders, criminal detention, etc.;
16. Subjects considered unsuitable for the study by the investigator for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to1year
  Assessed by the investigator according to RECIST V1.1
AEs | Up to 2 years
  AE, SAE, TRAE, irAE, AE leading to dose adjustment, AE leading to withdrawal from the trial, and laboratory data were summarized according to NCI-CTCAE V5.0

SECONDARY OUTCOMES:
Progression Free Survival | Up to 2 years
  Assessed by the investigator according to RECIST V1.1
Duration of Response | Up to 2 years
  Assessed by the investigator according to RECIST V1.1
Disease Control Rate | Up to 1 year
  Stable disease (SD) should persist for ≥6 weeks as assessed by the investigator according to RECIST V1.1
Overal Survival | Up to 2 years
  The estimation was based on Kaplan-Meier (KM) method

CONTACTS AND LOCATIONS:
Overall Officials: Overall Study Officials Xiaofeng, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
CRF
Supporting Information: CSR
Time Frame: 2022.8-2025.8
Access Criteria: CRF